CLINICAL TRIAL: NCT00963859
Title: Phase II Evaluation of Robotic-assisted Laparoscopic Extended Pelvic Lymph Node Dissection for Transitional Cell Carcinoma of the Bladder
Brief Title: Robotic-Assisted Laparoscopic Extended Pelvic Lymph Node Dissection for Transitional Cell Carcinoma of the Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0441
Record Dates: First submitted 2009-08-19; First posted 2009-08-24 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-04

CONDITIONS: Bladder Cancer
Keywords: Robotic-assisted laparoscopic surgery; Extended pelvic lymph node dissection; RA-PLND; Second-look open lymph node dissection; O-PLND; Radical Cystectomy; Urinary diversion; Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robotic-assisted laparoscopic surgery (Experimental): Robotic-assisted laparoscopic extended pelvic lymph node dissection
  Interventions: Procedure: Robotic-assisted laparoscopic surgery

INTERVENTIONS:
Procedure: Robotic-assisted laparoscopic surgery — During radical cystectomy, robotic-assisted technique used to perform cystectomy and pelvic lymph node dissections. Each patient will undergo a second-look open lymph node dissection once the incision is made at the end for the urinary diversion.

SUMMARY:
The goal of this clinical research study is to evaluate how many lymph nodes are left behind after robotic-assisted removal and are then found after a wider incision is made, in patients who are having their bladder removed for the treatment of bladder cancer.

The primary objective is to compare the lymph node yield achieved by performing a robotic-assisted laparoscopic extended pelvic lymph node dissection (RA-PLND) compared to a second-look open lymph node dissection (O-PLND) among patients undergoing radical cystectomy for transitional cell carcinoma of the bladder.

The secondary objectives will be to collect prospective outcomes data related to the performance of RA-PLND and robotic-assisted cystectomy (RA-C) including operative times, estimated blood loss, transfusions, complications, return to diet, utilization of pain medication, hospital length, return to regular activities.

DETAILED DESCRIPTION:
Study Background:

Research has shown that the more lymph nodes removed as part of a radical cystectomy (bladder removal) for invasive bladder cancer, the better. However, the number of lymph nodes removed varies from person to person. The standard surgical techniques such as robot-assisted procedures are new, and researchers want to be able to more reliably tell if the specific number of lymph nodes removed is enough to be considered a "complete" removal.

In this study, researchers will remove the required lymph nodes using a standard robotic-assisted procedure, and then remove any additional lymph nodes that remain and need to be removed, using a wider ("open") incision in the abdomen. This open technique is also being done for standard of care. It is needed in order to complete the "urinary diversion" part of the surgery (a procedure of surgically making way for urine to pass out of the body so that it does not go through the bladder).

The main goal of the study is to see if the robotic-assisted procedure removes all of the required lymph nodes. The open technique will allow researchers to evaluate how many lymph nodes were left behind after robotic-assisted removal.

It is possible that the machine may have problems and not be available for use on the scheduled day of surgery. If that happens, you will have the option to reschedule surgery or have standard open surgery. It is also possible that the machine could have problems during your surgery. If that happens, your doctor will continue with standard open surgery. Your study doctor will discuss these possible situations with you.

You will be asked to sign a separate consent form for these surgical procedures, which will describe the procedures and their risks in more detail.

Follow-up:

You will be asked to fill out a brief pain survey once a week for 7 weeks after surgery. The survey will take about 5 minutes to complete. You will also be given a diary to record your daily pain medication use. It will also take about 5 minutes to complete. You will continue to complete the questionnaire once a week and to fill out the diary daily for 6 weeks.

End-of-Study Visit:

You will visit the clinic 6-12 weeks after surgery for an end-of-study visit. You will have a chest x-ray. Your pain medication use and pain level surveys will be collected. After this visit, you will be off-study.

This is an investigational study. The robotic-assisted bladder removal is FDA approved for this purpose. Up to 60 patients will be enrolled in this study. All will be enrolled at The University of Texas (UT) MD Anderson Cancer Center (MDACC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are eligible for a radical cystectomy and who, in the opinion of the treating MDACC physician, are candidates for a robotic-assisted laparoscopic technique for management of the bladder and lymph nodes.
2. Diagnosis of transitional cell carcinoma of the bladder.
3. Medical fitness for open radical cystectomy by consensus of MDACC urology and anesthesia faculty (medicine/cardiology clearance by common best practice criteria).
4. Staging inclusion by cystoscopic biopsy and bimanual examination under anesthesia: carcinoma in-situ, T1, T2.

Exclusion Criteria:

1. Prior pelvic radiation.
2. Morbid obesity, i.e., body mass index (BMI)> 35.
3. Metastatic disease, bulky disease--T3a/b, prostatic stromal invasion.
4. Non-transitional cell histology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W. Davis, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Davis JW, Gaston K, Anderson R, Dinney CP, Grossman HB, Munsell MF, Kamat AM. Robot assisted extended pelvic lymphadenectomy at radical cystectomy: lymph node yield compared with second look open dissection. J Urol. 2011 Jan;185(1):79-83. doi: 10.1016/j.juro.2010.09.031. Epub 2010 Nov 12. PMID 21074799
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 10, 2007 to December 07, 2009; All recruitment done in a medical clinic setting.
Period: Overall Study
Arm/Group | Robotic-assisted Laparoscopic Surgery
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robotic-assisted Laparoscopic Surgery
Number analyzed (Participants) | 11
Age Continuous [Median (Full Range); unit: years] | 73 [40 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Median Yield of Robot Assisted and Second Look Open Pelvic Lymph Node Dissection to Compare the Lymph Node Yield Achieved
Description: The median yield (the lymph node count) allows for comparison of how many lymph nodes are left behind after robotic-assisted removal and are then found after a wider incision is made. Specifically a robot-assisted laparoscopic extended pelvic lymph node dissection (RA-PLND) is compared to a second-look open lymph node dissection (O-PLND) among participants undergoing radical cystectomy for urothelial carcinoma of the bladder. The median yield lymph nodes illustrate the adequacy of extended pelvic lymph node dissection using a robotic-assisted technique, i.e. whether the robotic-assisted laparoscopic radical cystectomy yields a sufficient number of lymph nodes to be oncologically equivalent to the open procedure.
Time Frame: 3 months including surgery and post-operative period.
Measure: Median (Full Range); unit: Nodes (Node Yield)
Arm/Group | Robotic-assisted Laparoscopic Surgery
Number analyzed (Participants) | 11
Nodes (Node Yield)
  RA-PLND | 43 [19 to 63]
  O-PLND | 4 [0 to 8]

2. Primary Outcome: Overall Percentage Median Yield
Description: The median yield (the lymph node count) allows for comparison of how many lymph nodes are left behind after robotic-assisted removal and are then found after a wider incision is made. Specifically a robot-assisted laparoscopic extended pelvic lymph node dissection (RA-PLND) is compared to a second-look open lymph node dissection (O-PLND) among participants undergoing radical cystectomy for urothelial carcinoma of the bladder. The median yield lymph nodes illustrates the adequacy of extended pelvic lymph node dissection using a robotic-assisted technique.
Time Frame: 3 months including surgery and post-operative period.
Measure: Number; unit: Percentage of Nodes (Node Yield)
Arm/Group | Robotic-assisted Laparoscopic Surgery
Number analyzed (Participants) | 11
Percentage of Nodes (Node Yield)
  RA-PLND | 93
  O-PLND | 7

ADVERSE EVENTS:
Time Frame: 20 months
Arm/Group | Robotic-assisted Laparoscopic Surgery
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Robotic-assisted Laparoscopic Surgery (N=11)
Bowel Leak (Surgical and medical procedures) | 1 — Bowel leak from the gastrointestinal anastomosis
Death (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Robotic-assisted Laparoscopic Surgery (N=11)
Ileus (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No